CLINICAL TRIAL: NCT04648358
Title: REDUCE Trial: The Effects of Perineural Dexamethasone on Scalp Nerve Blocks for Relief of Postcraniotomy Pain
Brief Title: REDUCE Trial: Perineural Dexamethasone on Scalp Nerve Blocks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Director of Department of Pain Management, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY 2018-034-02-9
Record Dates: First submitted 2020-11-22; First posted 2020-12-01 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Postoperative Pain; Craniotomy; Dexamethasone; Scalp Nerve Blocks
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): The control group will receive scalp nerve blocks with 0.5% bupivacaine, plus normal saline with epinephrine at 1:200,000
  Interventions: Drug: Bupivacaine
- DEX4mg group (Experimental): DEX4mg group will receive scalp nerve blocks with 0.5% bupivacaine, plus 4 mg dexamethasone with epinephrine at 1:200,000.
  Interventions: Drug: Dexamethasone combined with bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — The control group will receive scalp nerve blocks with 0.5% bupivacaine with epinephrine at 1:200,000, plus normal saline 1 ml. The anesthesiologist will perform scalp nerve blocks based on the group allocation 10 mins before the incision. Scalp nerve blocks will be performed according to the technique previously described by Pinosky et al.
  Arms: Control group
Drug: Dexamethasone combined with bupivacaine — The DEX4mg group will receive scalp nerve blocks with 0.5% bupivacaine with epinephrine at 1:200,000, plus 4 mg dexamethasone (1 ml). The anesthesiologist will perform scalp nerve blocks based on the group allocation 10 mins before the incision. Scalp nerve blocks will be performed according to the technique previously described by Pinosky et al.
  Arms: DEX4mg group

SUMMARY:
Pain is common in the first 2 days after major craniotomy. Inadequate analgesia may lead to an increased risk of postoperative complications. Most pain following craniotomy arises from the pericranial muscles and soft tissues of the scalp. Scalp nerve blocks with local anesthesia seem to provide effective, safe, however transient postoperative analgesia which does not seem to meet the requirements of craniotomy. Currently, peripheral dexamethasone has been observed to significantly prolong the duration of analgesia of nerve blocks (e.g., saphenous nerve block, adductor canal block, thoracic paravertebral block, brachial plexus nerve block). On the contrary, a study reported that perineural dexamethasone did not appear to prolong the analgesic time after supratentorial craniotomy. However, all patients in this study were given 24 mg of oral or intravenous dexamethasone regularly at least 7 days during the perioperative period, which possibly masked the role of single local low doses of perineural dexamethasone. Therefore, the analgesic effect of single dexamethasone for scalp nerve blocks without the backdrop of perioperative glucocorticoid deserves further clarification.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for elective supratentorial craniotomy under general anesthesia;
* age 18 to 64 years;
* an American Society of Anesthesiologists (ASA) physical status of I, II or III;
* preoperative Glasgow Coma Scale (GCS) score of 15/15.

Exclusion Criteria:

* History of chronic headache or chronic pain syndrome of any cause, psychiatric disorders, or uncontrolled epilepsy;
* Inability to understand or use the pain scales before surgery;
* Excessive alcohol or drug abuse, chronic opioid use (more than 2 weeks or 3 days per week for more than 1 month), use of drugs with confirmed or suspected sedative or analgesic effects, or use of any painkiller within 24 hours before surgery;
* Request of oral/intravenous glucocorticoid to decrease cerebral edema within 1 week before surgery;
* Pregnancy or breastfeeding;
* Extreme body mass index (BMI) (< 15 or > 35);
* Participation in another interventional trial that interferes with the intervention or outcome of this trial;
* Refusal or inability of the patient and/or legal guardian to provide informed consent;
* Coagulopathy;
* Infection around the puncture point;
* History of allergies to any of the study drugs.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 156 (Actual)
Dates: Start 2020-12-13 (Actual); Primary Completion 2023-01-02 (Actual); Study Completion 2023-01-02 (Actual)

PRIMARY OUTCOMES:
The duration of analgesia | Within 48 hours after surgery
  The time between the performance of the block and the administration of the first press the PCA demand button postoperatively.

SECONDARY OUTCOMES:
Sufentanil consumption | At 4, 12, 24 and 48 hours postoperatively
  The cumulative amount of sufentanil consumption by PCA
Numeric rating scale (NRS) | At 2, 4, 8, 12, 16, 20, 24, and 48 hours postoperatively
  NRS: 11-point scale in which 0 = no pain to 10 = worst imaginable pain. An NRS score ≥4 will be considered significant or moderate pain. An NRS score ≥7 will be considered severe pain. Meanwhile, the localization of the site of the pain will also be documented.
Glasgow Coma Scale (GCS) | At 2, 4, 8, 12, 16, 20, 24, and 48 hours postoperatively
  A scale for measuring level of consciousness, in which scoring is determined by three factors: amount of eye opening, verbal responsiveness, and motor responsiveness.
Postoperative nausea and vomiting (PONV) | Within 48 hours after surgery
  Vomiting will be defined as the forceful expulsion of gastric contents, and nausea will be defined as an unpleasant sensation associated with the urge to vomit.
Bradycardia | Within 48 hours after surgery
  Bradycardia will be defined as HR<60 beats/minute in at least two instances more than 5 minutes apart.
Hypotension | Within 48 hours after surgery
  Hypotension will be defined as any of the following: systolic BP <90 mm Hg for 5 minutes or a 35% decrease in mean arterial blood pressure.
Emergence delirium | Within 48 hours after surgery
  Emergence delirium will be assessed by the Sedation Agitation Scale (SAS), a 7-point scale on which a higher score represents greater agitation.
The length of stay (LOS) | About at 2 weeks after surgery
  The LOS will be defined as the number of nights spent in the hospital after surgery.
Patient satisfaction score (PSS) | At 2, 4, 8, 12, 16, 20, 24, and 48 hours postoperatively
  PSS: 0 for unsatisfactory to 10 for very satisfactory.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Flexman AM, Ng JL, Gelb AW. Acute and chronic pain following craniotomy. Curr Opin Anaesthesiol. 2010 Oct;23(5):551-7. doi: 10.1097/ACO.0b013e32833e15b9. PMID 20717011
- [Background] Dilmen OK, Akcil EF, Tunali Y, Karabulut ES, Bahar M, Altindas F, Vehid H, Yentur E. Postoperative analgesia for supratentorial craniotomy. Clin Neurol Neurosurg. 2016 Jul;146:90-5. doi: 10.1016/j.clineuro.2016.04.026. Epub 2016 May 4. PMID 27164511
- [Background] Pinosky ML, Fishman RL, Reeves ST, Harvey SC, Patel S, Palesch Y, Dorman BH. The effect of bupivacaine skull block on the hemodynamic response to craniotomy. Anesth Analg. 1996 Dec;83(6):1256-61. doi: 10.1097/00000539-199612000-00022. PMID 8942596
- [Background] Yang Y, Ou M, Zhou H, Tan L, Hu Y, Li Y, Zhu T. Effect of Scalp Nerve Block with Ropivacaine on Postoperative Pain in Patients Undergoing Craniotomy: A Randomized, Double Blinded Study. Sci Rep. 2020 Feb 13;10(1):2529. doi: 10.1038/s41598-020-59370-z. PMID 32054899
- [Background] Baloda R, Bhupal JP, Kumar P, Gandhi GS. Supraclavicular Brachial Plexus Block With or Without Dexamethasone as an Adjuvant to 0.5% Levobupivacaine: A Comparative Study. J Clin Diagn Res. 2016 Jun;10(6):UC09-12. doi: 10.7860/JCDR/2016/18325.8048. Epub 2016 Jun 1. PMID 27504384
- [Background] Jose R, Chakravarthy K, Nair S, Joseph M, Jeyaseelan V, Korula G. A Randomized Controlled Trial Studying the Role of Dexamethasone in Scalp Nerve Blocks for Supratentorial Craniotomy. J Neurosurg Anesthesiol. 2017 Apr;29(2):150-156. doi: 10.1097/ANA.0000000000000272. PMID 26756502
- [Derived] Zhao C, Jia Z, Shrestha N, Luo F. REDUCE trial: the effects of perineural dexamethasone on scalp nerve blocks for relief of postcraniotomy pain-a study protocol for a randomized controlled trial. Trials. 2021 Nov 4;22(1):772. doi: 10.1186/s13063-021-05747-y. PMID 34736497